CLINICAL TRIAL: NCT02189213
Title: Treatment of Pediatric Anxiety Disorders by Predicting Treatment Response Through Biocellular Markers and Sleep
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Insufficient funding
Sponsor: New York State Psychiatric Institute (Other)
Collaborators: Columbia University (Other)
Responsible Party: Principal Investigator, Amir A. Levine, Psychiatrist 2/Associate Professor of Clinical Psychiatry, New York State Psychiatric Institute
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 6884
Record Dates: First submitted 2014-07-07; First posted 2014-07-14 (Estimated); Results first posted 2021-10-11 (Actual); Last update posted 2021-10-11 (Actual); Status verified 2021-09

CONDITIONS: Generalized Anxiety Disorder; Separation Anxiety Disorder; Social Phobia
Keywords: anxiety; SSRI; biomarker; sleep; children; adolescents; young adults
MeSH Terms: conditions — Generalized Anxiety Disorder; Anxiety, Separation; Phobia, Social; Anxiety Disorders | interventions — Sertraline

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Sertraline (Active Comparator): Sertraline will be administered PO to treat anxiety disorders in children and adolescents. he following dosing schedules will be used: Sertraline will be titrated from 25mg once a day orally up to 200mg once a day orally, for 12 weeks. The titration will stop at the dose in which the participant shows a full response to the medication or experiences side effects that will inhibit titration.
  Interventions: Drug: Sertraline
- Control (No Intervention): There will be no intervention in this arm.

INTERVENTIONS:
Drug: Sertraline — Sertraline will be administered to treat anxiety disorders in children and adolescents.
  Other Names: Zoloft
  Arms: Sertraline

SUMMARY:
1 out of 8 children, adolescents, and young adults suffer from an anxiety disorder. Studies over the past decade show that selective serotonin-reuptake inhibitors (SSRIs), a class of medication that treats anxiety in adults, also works well in young adults, children, and adolescents with anxiety disorders, but only for about 50%. 50% will have undergone treatment for several months before it will be established that the medication is not working to treat the anxiety. The purpose of this study is to find a test that will predict treatment outcome from the beginning based on behavioral and biological measures.

DETAILED DESCRIPTION:
Current evidence based psychiatric treatment for child, adolescent, and young adult anxiety disorders involves a trial and error process. Pediatric psychiatrists start with the first line treatments (i.e. SSRI or psychotherapy), which requires from 4-8 weeks to work. There is a long interval between treatment initiation and response with only 50 to 60% likelihood that the treatment chosen will succeed in reducing anxiety symptoms. The science that will enable us to predict who will respond to medication treatment does not exist. Studies have demonstrated a correlation between cellular markers in white blood cells and psychiatric disorders suggesting that certain genes may also change their expression in peripheral cells in response to treatment of psychiatric disorders. Several studies report a significant decrease in expression of key genes that are involved in the pathophysiology of anxiety and depression in the brain, such as BDNF, CREB and HDAC5 levels in leukocytes of people with mood and anxiety disorders. The levels of BDNF, HDAC5 and CREB in white blood cells then respond to treatment and match that of controls after treatment with SSRIs. The increased accessibility to sequencing technology allows us to survey many more potential biomarkers than what was possible just several years ago. This may enable us to formulate a test that will predict, based on biocellular markers, treatment outcome in anxiety disorders for children, adolescents, and young adults before the onset of treatment. By finding molecular markers that can predict treatment success from the onset, the investigators can improve treatment outcomes considerably compared to current standard treatment practices. This kind of personalized medicine is the future of psychiatry.

ELIGIBILITY:
Inclusion Criteria:

1. Participants aged 8-25 years inclusive at the time of the consent/assent, either outpatient or inpatient if hospitalization is required for one of the following reasons:

   * It is presently unsafe for subject to stay at home because he/she may run away
   * Subject needs closer monitoring while being started on medications
   * Subject needs a level of care that is greater than once a week outpatient treatment and is willing to participate in the study.
2. Participant's parent or legally authorized representative (LAR) must provide signature of informed consent, and there must be documentation of assent by the participant.
3. Participant meets Diagnostic and Statistical Manual of Mental Disorders Fourth Edition (DSM-IV) or Fifth Edition (DSM-V) criteria for a clinically impairing anxiety disorder based on detailed psychiatric evaluation at screening including completion of the Anxiety Disorders Interview Schedule for DSM-IV or DSM-V Child Version (ADIS-C) and a Children's Global Assessment Scale (CGAS) score less than 65.
4. Participants who are female of child-bearing potential (defined as ≥9 years of age or if <9 years of age are post-menarchal) must have a negative urine pregnancy test at the Baseline Visit. Females of child-bearing potential must abstain from sexual activity that could result in pregnancy or agree to use acceptable methods of contraception. Condoms should be used with the following acceptable contraceptives:

   * Intrauterine devices,
   * Hormonal contraceptives (oral, depot, patch, injectable, or vaginal ring).
   * Other acceptable contraceptive methods are double barrier methods (e.g., condoms and diaphragms with spermicidal gel or foam).

Exclusion Criteria:

1. Participant has a current co-morbid psychiatric diagnosis of bipolar disorder, psychosis, a pervasive developmental disorder other than Asperger's Syndrome, an eating disorder, substance abuse disorder, or a sleep disorder of narcolepsy and/or sleep apnea.
2. Participant has any condition or illness which, in the opinion of the study doctor, represents as an inappropriate risk to the participant and/or could confound the interpretation of the study.
3. Participant has received any evidence-based psychosocial intervention in the past 6 weeks i.e. Individual Cognitive Behavioral Therapy, Group Cognitive Behavioral Therapy, or Social Effectiveness Training.
4. Participant is unwilling or unable to provide blood, urine, and/or saliva samples at designated visits.
5. Participant is female and is pregnant or is currently lactating.
6. Participant is currently considered at risk for suicide in the opinion of the study doctor, has made a suicide attempt within the past 6 months, or is currently reporting active suicidal ideation. Participants with intermittent passive suicidal ideation are not necessarily excluded based on the assessment of the study doctor. Control participants with any suicidal ideation will not be eligible for the study.
7. Participant has had a substance use disorder within the past 6 months.
8. Participant has a clinically important abnormality on drug and alcohol screen.
9. Participant has started or changed the dosage of medication (including herbal supplements) that has anxiolytic, anxiogenic, or central nervous system (CNS) effects within the past 3 months.
10. Participant has a known or suspected allergy, hypersensitivity, or clinically significant intolerance to any components found in the study drug.
11. Participant has had several failed attempts with SSRI treatment.
12. Participant has an acute illness and/or is taking short term medication at the time of initiation of the study.
13. Participant failed screening or was previously enrolled in this study
14. Participant is unable to read.

Ages: 8 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 14 (Actual)
Dates: Start 2014-07 (Actual); Primary Completion 2019-12 (Actual); Study Completion 2019-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Amir Levine, Principal Investigator — New York State Psychiatric Institue
Locations (1):
- NYSPI, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Sertraline: Sertraline was administered PO to treat anxiety disorders in children and adolescents. One of the following dosing schedules will be used:
  Sertraline will be titrated from 25mg once a day orally up to 200mg once a day orally, for 12 weeks, or, the titration was stopped at the dose in which the participant shows a full response to the medication or experiences side effects that will inhibit titration.
- Healthy Control: Healthy control will not be treated.
Period: Overall Study
Arm/Group | Sertraline | Healthy Control
Started | 13 | 1
Completed | 7 | 1
Not Completed | 6 | 0

BASELINE CHARACTERISTICS:
Groups:
- Sertraline: Sertraline will be administered PO to treat anxiety disorders in children and adolescents. One of the following dosing schedules will be used:
  Sertraline will be titrated from 25mg once a day orally up to 200mg once a day orally, for 12 weeks, or the titration will stop at the dose in which the participant shows a full response to the medication or experiences side effects that will inhibit titration.
- Total: Total of all reporting groups
Arm/Group | Sertraline | Control | Total
Number analyzed (Participants) | 13 | 1 | 14
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 12 | 0 | 12
  Between 18 and 65 years | 1 | 1 | 2
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 1 | 9
  Male | 5 | 0 | 5
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 1 | 3
  White | 11 | 0 | 11
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 13 | 1 | 14

OUTCOME MEASURES:

1. Primary Outcome: Clinical Global Impression-Improvement (CGI-I) Score
Description: The CGI-I score at the final visit will determine treatment response.
  The CGI-Improvement scale comprises a one-item measures evaluating the following change from the initiation of treatment on a seven-point scale.
  The following one query is rated on a seven-point scale: "Compared to the patient's condition at admission to the project [prior to medication initiation], this patient's condition is: 1=very much improved since the initiation of treatment; 2=much improved; 3=minimally improved; 4=no change from baseline (the initiation of treatment); 5=minimally worse; 6= much worse; 7=very much worse since the initiation of treatment.
  CGI-I scale of 1-2 is considered response to treatment. Anything below that is considered non-response to sertraline treatment.
Time Frame: Final visit, at 12 weeks of treatment
Population: There were two males and two females in the responder group and two females and one male in the non-responder group.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Sertraline Responders: Responders will have either a score of 1 or 2 on the Clinical Global Impressions (CGI) Improvement Scale. The CGI-Improvement scale comprises a one-item measures evaluating the following change from the initiation of treatment on a seven-point scale.
  The following one query is rated on a seven-point scale: "Compared to the patient's condition at admission to the project [prior to medication initiation], this patient's condition is: 1=very much improved since the initiation of treatment; 2=much improved; 3=minimally improved; 4=no change from baseline (the initiation of treatment); 5=minimally worse; 6= much worse; 7=very much worse since the initiation of treatment.
  CGI-I scale of 1-2 is considered response to treatment. Anything below that is considered non-response to sertraline treatment.
- Sertraline Non-Responders: Non-Responders will have a score of 3 or greater than 3 on the Clinical Global Impressions (CGI) Improvement Scale. The CGI-Improvement scale comprises a one-item measures evaluating the following change from the initiation of treatment on a seven-point scale.
  The following one query is rated on a seven-point scale: "Compared to the patient's condition at admission to the project [prior to medication initiation], this patient's condition is: 1=very much improved since the initiation of treatment; 2=much improved; 3=minimally improved; 4=no change from baseline (the initiation of treatment); 5=minimally worse; 6= much worse; 7=very much worse since the initiation of treatment.
  CGI-I scale of 1-2 is considered response to treatment. Anything below that is considered non-response to sertraline treatment.
Arm/Group | Sertraline Responders | Sertraline Non-Responders
Number analyzed (Participants) | 4 | 3
units on a scale | 1.00 (1.40) | 3.66 (2.12)
Statistical Analysis 1: Comparison: Sertraline Responders vs Sertraline Non-Responders; At least 50% of subjects will respond to Sertraline treatment (CGI greater than or equal to 2); Test type: Other — The parameters were the CGI-Improvement scale which comprises a one-item measures evaluating the following change from the initiation of treatment on a seven-point scale. The hypothesis is that ~50% of subjects receiving treatment will not respond; p = 0.0002, t-test, 2 sided

ADVERSE EVENTS:
Time Frame: Adverse event data was collected for 12 weeks during the duration the patients were receiving medications. Only participants who were treated and healthy controls were monitored/assessed for adverse events.
Description: We collected adverse events using the Pediatric Adverse Event Rating Scale (PAERS-Clinician)
Arm/Group | Sertraline | Healthy Control
All-Cause Mortality (participants affected / at risk) | 0/8 | 0/1
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/1
Other Adverse Events (participants affected / at risk) | 0/8 | 0/1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2020-05-15): https://cdn.clinicaltrials.gov/large-docs/13/NCT02189213/Prot_000.pdf
  • Statistical Analysis Plan (2021-08-30): https://cdn.clinicaltrials.gov/large-docs/13/NCT02189213/SAP_001.pdf